CLINICAL TRIAL: NCT04462640
Title: Management of Infant Digestive Disorders and Quality of Life
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Keyrus Biopharma (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A03340-57
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Infant Nutrition Disorders; Gastrointestinal Dysfunction
Keywords: Quality of life; Infants; Regurgitation; Colic
MeSH Terms: conditions — Infant Nutrition Disorders; Gastroesophageal Reflux; Colic | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- regurgitation: 45 infants aged 0 to 5 months suffering from regurgitation
  Interventions: Other: Management of Infant Digestive Disorders and Quality of Life
- colic: 45 infants aged 0 to 5 months suffering from colic
  Interventions: Other: Management of Infant Digestive Disorders and Quality of Life

INTERVENTIONS:
Other: Management of Infant Digestive Disorders and Quality of Life — The variation of the QUALIN score on D30 compared to inclusion (D0) will be described and compared using a Student test for paired data in the case of a normal distribution or a test of the ranks signed by Wilcoxon otherwise.

SUMMARY:
The objective of the study is to measure the evolution of the quality of life in infants between 0 and 5 months old, not breastfed and suffering from regurgitation or colic.

DETAILED DESCRIPTION:
The objective of the study is to measure the evolution of the quality of life in infants between 0 and 5 months old, not breastfed and suffering from regurgitation or colic, following nutritional management of these disorders by a preparation for thickened infants, reduced in lactose content and supplemented with Lactobacillus reuteri DSM 17938. Quality of life is assessed using the QUALIN questionnaire

ELIGIBILITY:
Inclusion Criteria:

Full-term infants (> 37 weeks gestation and <42 weeks gestation), less than 4 months of age at recruitment

* Infants with regurgitation and / or colic defined according to Rome IV criteria
* Non-breastfed infants
* Parents who understand and speak French fluently
* Parents agreeing to send their email address and having a computer tool (computer, tablet or smartphone) allowing them to complete the QoL questionnaires and the satisfaction questionnaire
* Parents having understood the protocol and the information given and having given the participation agreement including their acceptance to return for consultation with the same doctor after a period of 30 days.

Exclusion Criteria:

Infant born prematurely (<37 weeks)

• Intercurrent pathology other than a functional intestinal disorder which can by themselves cause, directly or as a result of treatments, a functional intestinal disorder: Study Management of infant digestive disorders and Quality of life

* Food allergy
* Digestive pathology (Gastroenteritis, celiac disease, high or low digestive malformations….)
* Heart failure, cyanogenic heart disease
* Chronic respiratory diseases (bronchopulmonary dysplasia, malformations, respiratory failure)
* Neurological pathologies (Cerebral palsy, intracranial hypertension, convulsive state)
* Congenital metabolic pathologies
* Genetic diseases
* Kidney malformations, Vesicoureteral reflux, Kidney failure.
* Drug treatment in progress and which will be continued during the study, other than vitamins (D, K, ...)
* Partial or total breastfeeding
* Infants already fed:
* with a hypoallergenic formula (HA)
* or with a high hydrolyzate of cow's milk proteins or formula based on rice protein hydrolyzate
* Growth retardation (weight and or height less than or equal to - 2 DS) or break in the weight curve (no weight gain or weight loss in the past month) Prescription of drugs or food supplements other than vitamins at the end of the visit

Ages: 1 Week to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants between 0 and 5 months
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Quality of life in infants with regurgitation and colic | 4 months
  The main endpoint will be an increase in the QUALIN (QUALIté de vie du Nourrison) score on D30 compared to inclusion (D0) according to the 2 groups of patients: regurgitation only and colic only. This score is between -68 to +68. An increase in score means an improvement in symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sandra Brancato, Brignon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chouraqui JP, Brancato S, Delmas B, Hanh T. Effectiveness of a starch thickened infant formula with reduced lactose content, probiotics and prebiotics on quality of life and clinical outcome in infants with regurgitation and/or colic. Front Nutr. 2023 May 25;10:1164722. doi: 10.3389/fnut.2023.1164722. eCollection 2023. PMID 37305080